CLINICAL TRIAL: NCT07077473
Title: A Retrospective Study Observing the Efficacy and Safety of Different Drugs Used in Real-world Familial Mediterranean Fever (FMF) Cases
Brief Title: Observing the Efficacy and Safety of Different Drugs Used in Real-world Familial Mediterranean Fever (FMF) Cases
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Pfizer (Industry); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, YIKAI YU, Doctor, Tongji Hospital
Other Study IDs: TJ-IRB202412016
Record Dates: First submitted 2025-06-21; First posted 2025-07-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Familial Mediterranean Fever (FMF )
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: real word drugs — real word drugs

SUMMARY:
retrospective observe the efficacy and safety of different drugs used in familial Mediterranean fever (FMF) cases in real-world

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Familial Mediterranean fever (FMF) patients (Tel Hashomer criteria)

Exclusion Criteria:

* Have a history of mental illness, or alcohol and drug dependence；
* Pregnant, with severe infection, severe cardiac insufficiency, severe liver or kidney dysfunction；
* Complicated with tumors, organ transplants, etc. which have significant impact on the immune system or require the use of immunosuppressants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: familial Mediterranean fever (FMF) patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical responses graded as Patient Global Assessment (PGA ) decrease | From baseline,4, 8, 12, 24 and week 52
  The treatment outcome was graded as PGA decrease:in-response, partial response, good response, or clinical remission corresponding to symptomatic improvement <30%, 30% to 50%, 50% to 70%, or >70%, respectively. PGA is a subjective measure where patients rate their overall disease activity or health status on a scale like a visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No